CLINICAL TRIAL: NCT05746442
Title: Ending Tobacco Use Through Interactive Tailored Messaging for Cambodian People Living With HIV/AIDS (Project END-IT)
Brief Title: Ending Tobacco Use Through Interactive Tailored Messaging for Cambodian People Living With HIV/AIDS
Acronym: ProjectENDIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Oklahoma (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCC-21528; U01CA261598 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; HIV
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (Active Comparator): Participants will receive brief advice and education materials to quit smoking along with brief weekly assessments to be completed on a smartphone. They will also receive a 8 week supply of of nicotine replacement therapy in the form of nicotine patches.
  Interventions: Drug: Nicotine patch; Behavioral: Brief Advice to Quit and Smoking Cessation Self Help Materials; Behavioral: Diet Assessment
- Automated Messaging Treatment Group (Experimental): Participants will receive brief advice and education materials to quit smoking, along with brief weekly assessments and an interactive phone-based treatment program delivered on a smartphone. They will also receive a 8 week supply of of nicotine replacement therapy in the form of nicotine patches.
  Interventions: Behavioral: Smartphone-delivered Automated Messaging; Drug: Nicotine patch; Behavioral: Brief Advice to Quit and Smoking Cessation Self Help Materials

INTERVENTIONS:
Behavioral: Smartphone-delivered Automated Messaging — An interactive smartphone based intervention will provide weekly smoking-related assessments and personalized automated messages designed to increase motivation, self-efficacy, use of coping skills, social support and to reduce nicotine withdrawal symptoms and stress for a 26 week period.
  Arms: Automated Messaging Treatment Group
Drug: Nicotine patch — Participants will be provided with a 8 week supply of nicotine patches
Behavioral: Brief Advice to Quit and Smoking Cessation Self Help Materials — Participants will receive self-help materials from Khmer Quit Now, a national smoking cessation campaign in Cambodia
Behavioral: Diet Assessment — Participants will be asked to complete brief weekly smartphone assessments about their diet for a 26-week period
  Arms: Standard Care Group

SUMMARY:
The goal of this research study is to test how well an automated text messaging smoking treatment program helps smokers with HIV quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* 1) being aged ≥18 years
* 2) being HIV-positive
* 3) self-reporting as a current combustible cigarette smoker (smoked ≥100 cigarettes in lifetime and currently smoke ≥1 cigarettes/day)
* 4) willing to set a date for a quit attempt within 2 weeks of study enrollment
* 5) being able to provide written informed consent to participate
* 6) being able to read Khmer (score ≥4 points on the Rapid Estimate of Adult Literacy in Medicine-Short Form

Exclusion Criteria:

* 1) history of a medical condition that precludes use of nicotine replacement therapy
* 2) physician/clinician deemed ineligible to participate based on medical or psychiatric condition
* 3) enrolled in another cessation program or use of other cessation medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Self Reported 7 Day Abstinence Smoking Status | 12 Month Follow-Up
  Participants will self report 7-day abstinence smoking status
Smoking Status by Expired Carbon Monoxide | 12 Month Follow-up
  Investigators will use a CO monitor to verify smoking status biochemically

SECONDARY OUTCOMES:
Self Reported 7 Day Abstinence Smoking Status at 3 Months | At 3 Months
  Participants will self report 7-day abstinence smoking status
Smoking Status by Expired Carbon Monoxide at 3 Months | At 3 Months
  Investigators will use a CO monitor to verify smoking status biochemically
Self Reported 7 Day Abstinence Smoking Status at 6 Months | At 6 Months
  Participants will self report 7-day abstinence smoking status
Smoking Status by Expired Carbon Monoxide at 6 Months | At 6 Months
  Investigators will use a CO monitor to verify smoking status biochemically

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, Dr.PH, Principal Investigator — Moffitt Cancer Center; Thanh Bui, Dr.PH, Principal Investigator — Phnom Penh
Locations (3):
- Cambodia (3):
  - National AIDS Authority, Phnom Penh
  - National Center for HIV/AIDS, Dermatology and STD, Phnom Penh
  - National Institute of Public Health, Phnom Penh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bui TC, Hoogland CE, Chhea C, Sopheab H, Ouk V, Samreth S, Hor B, Vidrine JI, Businelle MS, Shih YCT, Sutton SK, Jones SR, Shorey Fennell B, Cottrell-Daniels C, Frank-Pearce SG, Ngor C, Kulkarni S, Vidrine DJ. Ending Tobacco Use Through Interactive Tailored Messaging for Cambodian People With HIV (Project EndIT): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 29;12:e48923. doi: 10.2196/48923. PMID 37384390